CLINICAL TRIAL: NCT05400837
Title: Patient Centered Mobile Health Technology Enabled Atrial Fibrillation Management: A Pilot Randomized Clinical Trial
Brief Title: Patient Centered Mobile Health Technology Enabled Atrial Fibrillation Management
Acronym: mTECHAFib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00321575
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation; Behavior
Keywords: Remote Patient Monitoring; Atrial Fibrillation; Risk Factor Modification; Digital Health; Mobile Health
MeSH Terms: conditions — Atrial Fibrillation; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Corrie Virtual Atrial Fibrillation Management Program (Experimental): Multicomponent virtual atrial fibrillation management program
  Interventions: Combination Product: Corrie Virtual Atrial Fibrillation Management Program
- Usual Care (No Intervention): Receives usual care. Usual care is defined as care according to the patients care team's standard practice

INTERVENTIONS:
Combination Product: Corrie Virtual Atrial Fibrillation Management Program — Intervention aims to implement guideline-recommended Afib care
  Arms: Corrie Virtual Atrial Fibrillation Management Program

SUMMARY:
The overall objective of this proposal is to evaluate the feasibility of a comprehensive digital atrial fibrillation (AFib) management tool that will empower patients to a) take an active role in learning about AFib management options, starting and adhering to evidence-based therapies and lifestyle changes and b) to guide the patients during AFib episodes which are associated with anxiety and impairment in quality of life.

Researchers plan to evaluate the feasibility and preliminary efficacy of this novel digital toolkit in improving quality of life and decreasing AFib burden in a pilot randomized clinical trial (RCT).

ELIGIBILITY:
Inclusion Criteria

* 18 years or older
* Non- valvular Paroxysmal Atrial Fibrillation

Exclusion Criteria

* Non-English speaking
* Has previously been evaluated by a cardiologist or electrophysiologist
* Mitral Stenosis
* Presence of Artificial Heart Valve
* Severe valvular disease (any)
* Physical disability that would preclude technology use, safe and adequate exercise performance
* Hearing or Visual Impairment that would preclude technology use
* History of fall one or more times in the last year
* Hypertrophic obstructive cardiomyopathy with peak resting left ventricular outflow gradient of >25 mmHg
* Known aortic dissection
* Severe resting arterial hypertension (SBP >200 mmHg or diastolic BP >110mmHg) upon enrollment (obtained during clinic visit)
* Mental impairment leading to inability to cooperate with study procedures
* Untreated high degree atrioventricular block
* Atrial fibrillation with rapid ventricular rate (Resting heart rate at enrollment visit >110) upon enrollment (obtained during clinic visit)
* History of cardiac arrest, sudden death
* MI or cardiac surgery complications of cardiogenic shock and/or congestive heart failure (CHF) and/or signs/symptoms of post-procedure ischemia
* Left ventricular ejection fraction <40%
* Clinically significant depression
* Presence of implanted cardiac device
* Incomplete revascularization procedure
* Pregnancy
* Previous open-heart surgery
* Unsafe to participate in the program as per treating clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spragg, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from outpatient electrophysiology clinics at Johns Hopkins Hospital. A study coordinator reviewed EMRs and let clinicians know which patients were eligible. The clinician introduced the patient to the study, and if they were interested, the study coordinator talked to the patient after their appointment. Interested patients signed informed consent, were randomized, and onboarded to the study the same day.
Pre-assignment Details: Participants were assigned their group immediately after signing consent.
Period: Overall Study
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Started | 30 | 31
Completed | 25 | 29
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Population: Data was excluded for one participant who asked to have their data deleted from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Data was excluded for one participant who asked to have their data deleted from the study.
  years | 65 [58.25 to 70.5] | 69 [63.25 to 71.75] | 67.5 [60 to 71.25]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data was excluded for one participant who asked to have their data deleted from the study.
  Participants
    Female | 10 | 13 | 23
    Male | 20 | 17 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data was excluded for one participant who asked to have their data deleted from the study.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 2 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 0 | 2
    White | 26 | 28 | 54
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0
Quality of life as assessed by the Atrial Fibrillation Effect on Quality-of-Life [Mean (Standard Deviation); unit: Survey score] — Measured by Atrial Fibrillation Effect on Quality-of-Life (AFEQT), which consists of 20 items. Score ranges from 0 to 100 with higher scores signifying better quality of life. Population: Some participants chose not to complete this questionnaire.
  Survey score
    number analyzed (Participants) | 23 | 29 | 52
    (all) | 78.7 (24.1) | 73.1 (31.1) | 75.6 (28.0)
Atrial Fibrillation (AF) Severity as assessed by the Atrial Fibrillation Severity Scale [Mean (Standard Deviation); unit: Survey score] — Measured by the Atrial Fibrillation Severity Scale (AFSS) - validated 19 item questionnaire. Includes 5 subscores. AF burden is the sum of AF duration, AF severity, and AF frequency, and ranges from 3 to 30, with 30 being highest burden. AF duration, severity, and frequency each range from 1 to 10. The final subscore is AF symptoms, which ranges from 0-35 with 35 indicating worst possible symptoms. Population: Some participants chose not to complete this questionnaire
  Survey score
    AF burden subscore: number analyzed (Participants) | 23 | 29 | 52
    AF burden subscore | 12.8 (5.4) | 13.2 (3.7) | 13.0 (4.5)
    AF duration subscore: number analyzed (Participants) | 23 | 30 | 53
    AF duration subscore | 4.1 (2.8) | 4.3 (2.1) | 4.2 (2.4)
    AF severity subscore: number analyzed (Participants) | 23 | 30 | 53
    AF severity subscore | 5.3 (2.7) | 5.4 (2.3) | 5.4 (2.5)
    AF frequency subscore: number analyzed (Participants) | 23 | 30 | 53
    AF frequency subscore | 3.0 (3.0) | 3.4 (1.8) | 3.2 (2.5)
    AF symptoms subscore: number analyzed (Participants) | 23 | 30 | 53
    AF symptoms subscore | 6.3 (5.3) | 7.9 (6.5) | 7.2 (6.0)
Skills in applying electronic health information to health problems [Mean (Standard Deviation); unit: Survey score] — Measured by 10-item questionnaire eHealth Literacy Scale. Scores range from 10-50 with a higher score indicating higher electronic health information literacy. Population: Some participants chose not to complete this questionnaire
  Survey score
    number analyzed (Participants) | 23 | 30 | 53
    (all) | 38.2 (4.8) | 40.2 (4.9) | 39.3 (4.9)
Depressive symptoms as assessed by the Patient Health Questionnaire 8 [Mean (Standard Deviation); unit: Survey score] — Measured by Patient Health Questionnaire 8 (PHQ - 8) - 8-item measure with (≤4: no depressive symptom, 5-9: mild, ≥10: moderate to severe depressive symptoms). Score range 0-27, higher score more depressive symptoms. Population: Some participants chose not to complete this questionnaire
  Survey score
    number analyzed (Participants) | 21 | 30 | 51
    (all) | 1.0 (5.0) | 2.0 (5.0) | 1.6 (5.0)
Anxiety as assessed by the Generalized Anxiety Disorder 7 score [Mean (Standard Deviation); unit: Survey score] — Generalized Anxiety Disorder 7 (GAD 7) - score ranges from 0 to 21 with higher scores indicating more anxiety. Population: Some participants chose not to complete this questionnaire
  Survey score
    number analyzed (Participants) | 23 | 30 | 53
    (all) | 0 (4.0) | 2.0 (4.0) | 1.1 (4.0)
Stress level as assessed by the Perceived Stress Score [Mean (Standard Deviation); unit: Survey score] — Measured by Perceived Stress Score (PSS-10), 10 item questionnaire where score ranges from 0-40 with higher scores indicating higher level of stress. Population: Some participants chose not to complete this questionnaire
  Survey score
    number analyzed (Participants) | 21 | 30 | 51
    (all) | 10.1 (5.1) | 10.0 (13.0) | 10.0 (9.5)
Alcohol use as assessed by the Alcohol Use Disorders Identification Test [Mean (Standard Deviation); unit: Survey score] — As assessed by The Alcohol Use Disorders Identification Test (AUDIT), 10-item questionnaire. The score range is from 0 to 40 with 0 referring to abstainer with no history of alcohol abuse and higher scores indicate gradually higher and hazardous alcohol dependence. Population: Some participants chose not to complete this questionnaire
  Survey score
    number analyzed (Participants) | 23 | 30 | 53
    (all) | 2.0 (2.5) | 2.0 (3.0) | 2.0 (2.8)
Physical Activity as assessed by the Rapid Assessment of Physical Activity [Mean (Standard Deviation); unit: Survey score] — Physical Activity will be assessed by The Rapid Assessment of Physical Activity (RAPA). Part 1 is scored from 1 to 5 where 5 is the optimal level of physical activity, and 1 is completely sedentary. Part 2 measures flexibility/calisthenics exercise frequency and is scored from 0-3 where 3 is optimal. Population: Some participants chose not to complete this questionnaire
  Survey score
    RAPA Part 1 score: number analyzed (Participants) | 23 | 30 | 53
    RAPA Part 1 score | 5.0 (1.0) | 5.0 (1.0) | 5.0 (1.0)
    RAPA Part 2 score: number analyzed (Participants) | 23 | 30 | 53
    RAPA Part 2 score | 1.0 (2.0) | 2.0 (3.0) | 1.6 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Continue Study Participation at 12 Weeks
Description: Feasibility assessed by retention at 12 weeks (number of individuals who continue study participation (defined by App interaction, Coaching call participation or follow up survey completion)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 30 | 31
Participants | 26 | 29

2. Secondary Outcome: Quality of Life as Assessed by the Atrial Fibrillation Effect on Quality-of-Life
Description: Measured by Atrial Fibrillation Effect on Quality-of-Life (AFEQT), which consists of 20 items. Score ranges from 0 to 100 with higher scores signifying better quality of life.
Time Frame: 12 weeks
Population: Some participants chose not to complete this survey.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 23 | 29
score on a scale | 87.0 (24.1) | 76.0 (31.5)

3. Secondary Outcome: Atrial Fibrillation (AF) Severity as Assessed by the Atrial Fibrillation Severity Scale
Description: Measured by the Atrial Fibrillation Severity Scale (AFSS) - validated 19 item questionnaire. Includes 5 subscores. AF burden is the sum of AF duration, AF severity, and AF frequency, and ranges from 3 to 30, with 30 being highest burden. AF duration, severity, and frequency each range from 1 to 10. The final subscore is AF symptoms, which ranges from 0-35 with 35 indicating worst possible symptoms.
Time Frame: 12 weeks
Population: Some participants chose not to complete this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 23 | 29
score on a scale
  AF burden score (sum of duration, severity, and frequency subscores) | 11.3 (4.5) | 12.7 (5.0)
  AF duration score | 3.1 (2.4) | 4.3 (2.7)
  AF severity score | 4.6 (2.8) | 5.4 (2.6)
  AF frequency score | 3.6 (2.5) | 3.0 (1.7)
  AF symptoms score | 3.0 (4.0) | 7.6 (7.8)

4. Secondary Outcome: Skills in Applying Electronic Health Information to Health Problems
Description: Measured by 8-item questionnaire eHealth Literacy Scale. Scores range from 10-50 with a higher score indicating higher electronic health literacy.
Time Frame: 12 weeks
Population: Some participants chose not to complete this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 23 | 29
score on a scale | 40.0 (4.0) | 40.1 (5.6)

5. Secondary Outcome: Depressive Symptoms as Assessed by the Patient Health Questionnaire 8
Description: Measured by Patient Health Questionnaire 8 (PHQ - 8) - 8-item measure with (≤4: no depressive symptom, 5-9: mild, ≥10: moderate to severe depressive symptoms). Score range 0-27 with higher score indicating more depressive symptoms.
Time Frame: 12 weeks
Population: Some participants chose not to complete this survey
Measure: Mean (Standard Deviation); unit: Survey score
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 21 | 29
Survey score | 1.0 (4.0) | 3.0 (3.0)

6. Secondary Outcome: Anxiety as Assessed by the Generalized Anxiety Disorder 7 Score
Description: Generalized Anxiety Disorder 7 (GAD 7) - score ranges from 0 to 21 with higher scores indicating more anxiety.
Time Frame: 12 weeks
Population: Some participants chose not to complete this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 23 | 29
score on a scale | 1.0 (2.0) | 1.0 (3.0)

7. Secondary Outcome: Stress Level as Assessed by the Perceived Stress Score
Description: Measured by Perceived Stress Score (PSS-10), 10 item questionnaire where score ranges from 0-40 with higher scores indicating higher level of stress.
Time Frame: 12 weeks
Population: Some participants chose not to complete this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 23 | 29
score on a scale | 10.1 (5.1) | 11.5 (8.1)

8. Secondary Outcome: Physical Activity as Assessed by the Rapid Assessment of Physical Activity
Description: Physical Activity will be assessed by The Rapid Assessment of Physical Activity (RAPA). Part 1 scores range from 1-5 with increasing scores indicating higher levels of activity, 5 being optimal. Part 2 is scored from 0-3 and measures the amount of flexibility and calisthenics exercise a person completes, with 3 being optimal.
Time Frame: 12 weeks
Population: Some participants chose not to complete this survey
Measure: Mean (Standard Deviation); unit: Survey score
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 23 | 29
Survey score
  RAPA Part 1 score | 5.0 (0.5) | 5.0 (1.0)
  RAPA Part 2 score | 1.0 (2.0) | 2.0 (3.0)

9. Secondary Outcome: Alcohol Use as Assessed by the Alcohol Use Disorders Identification Test
Description: As assessed by The Alcohol Use Disorders Identification Test (AUDIT), 10-item questionnaire. The score range is from 0 to 40 with 0 referring to abstainer with no history of alcohol abuse and higher scores indicate gradually higher and hazardous alcohol dependence.
Time Frame: 12 weeks
Population: Some participants chose not to complete this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 23 | 29
score on a scale | 2.0 (2.0) | 2.0 (3.0)

10. Secondary Outcome: Diet as Assessed by the Rate Your Plate (RYP) Scale
Description: Measured by Rate Your Plate (RYP) scale. A 27 item scale administered at 12 weeks with the following scoring system: Score ranges from 27-81.
  Score of 27-45: There are many ways you can make your eating habits healthier. 46-63: There are some ways you can make your eating habits healthier. 64-81: Higher score indicates participant is making many healthy choices.
Time Frame: 12 weeks
Population: Some participants chose not to complete this survey
Measure: Mean (Standard Deviation); unit: Survey score
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 23 | 29
Survey score | 65.1 (5.3) | 64.0 (6.2)

11. Secondary Outcome: Blood Pressure
Description: Measured in millimeters of mercury (mmHg).
Time Frame: 12 weeks
Population: Some participants did not complete the 12-week follow-up visit where blood pressure was assessed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 24 | 28
mmHg
  Systolic blood pressure | 123.1 (16.3) | 123.3 (14.2)
  Diastolic blood pressure | 75.6 (8.7) | 73.4 (9.9)

12. Secondary Outcome: Body Mass Index (BMI)
Description: Measured in kilograms over meter squared (Kg/m^2).
Time Frame: 12 weeks
Population: Not all participants completed the 12-week follow-up visit where weight was measured.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 24 | 29
kg/m^2 | 29.6 (4.8) | 29.9 (7.0)

13. Secondary Outcome: Satisfaction With Intervention
Description: Measured by the System Usability Scale (SUS), modified for the intervention. The SUS score ranges from 0-100, where 0 is "worst imaginable" and 100 is "best imaginable." The average score is 68.0, a good score is between 71.4-85.4. 85.5 and above is considered excellent. Higher score more satisfaction.
Time Frame: 12 weeks
Population: Participants in usual care did not receive intervention and so did not rate their satisfaction. Not all participants in the intervention chose to complete the survey.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 20 | 0
score on a scale | 78.25 [70.5 to 86.75] |

14. Other Pre Specified Outcome: At-home Sleep Study Results
Description: Patients completed an at-home sleep study and received a diagnosis of no sleep apnea, mild sleep apnea, moderate sleep apnea, or severe sleep apnea, based on their AHI (apnea-hypopnea index). AHI is measured in breathing disturbance events per hour. An AHI <5 indicates no sleep apnea, from 5-15 is mild, 16-30 is moderate, and >30 is severe sleep apnea.
Time Frame: Studies were completed one time between enrollment and end of treatment at 12 weeks
Population: The control group did not complete a sleep study. Not all members of the intervention group chose to complete the sleep study.
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
Number analyzed (Participants) | 26 | 0
Participants
  Diagnosed with mild sleep apnea | 4 | 0
  Diagnosed with moderate to severe sleep apnea | 8 | 0
  Not diagnosed with sleep apnea | 14 | 0

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 12 weeks
Description: The investigators asked participants to report any adverse events up to the end of follow-up (12 weeks). Adverse events were adjudicated by the principal investigator.
Arm/Group | Corrie Virtual Atrial Fibrillation Management Program | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/31
Other Adverse Events (participants affected / at risk) | 4/30 | 5/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corrie Virtual Atrial Fibrillation Management Program (N=30) | Usual Care (N=31)
Pulmonary embolism (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corrie Virtual Atrial Fibrillation Management Program (N=30) | Usual Care (N=31)
Hospitalization (General disorders) | 2 (2) | 2 (2)
Emergency department visit (General disorders) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT05400837/Prot_SAP_000.pdf